CLINICAL TRIAL: NCT01774760
Title: Reproducibility of Intratumor Distribution of 18F-EF5 in Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Heikki Minn, Professor, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T14/2013
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: 18F-EF5; PET/CT; Reproducibility
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

ARMS (1):
- Patients with stage III-IV head and neck cancer (Experimental): 18F-EF5 PET/CT scan
  Interventions: Drug: 18F-EF5; Procedure: Pretreatment PET/CT-scan (performed two times)

INTERVENTIONS:
Drug: 18F-EF5
  Other Names: PET/CT static imaging
Procedure: Pretreatment PET/CT-scan (performed two times)

SUMMARY:
The results of previous studies suggest further development of [18F]EF5 as a PET tracer for imaging hypoxia. This is a non-randomized prospective study to obtain information on reproducibility of [18F]EF5 intratumor distribution using repeated pretreatment PET/CT scans.

DETAILED DESCRIPTION:
All patients will undergo normal diagnostic and staging procedures, including a conventional 18F-FDG PET/CT scan for the purpose of RT or surgical planning. In addition to that, an 18F-EF5 PET/CT scan will be performed on a separate day. The patients receive intravenous injection of 250-350 MBq of [18F]EF5. After that, a venous blood sample will be obtained for measurement of plasma radioactivity. A low-dose CT (helical) will be performed for attenuation correction and anatomical reference. After that, a PET scan will be performed (starting at 3 h after injection). The second 18F-EF5 scan will be performed in a similar way 4-7 days after the first scan. A representative histologic sample of primary tumor is pre-condition for study and an effort is made to store part of fresh histologic material in liquid nitrogen for later use in immunohistochemical analysis.

Patients are scheduled to undergo preoperative or definitive chemoradiotherapy using current clinical standards after completion of the current protocol. Follow-up information (event-free survival and overall survival) will be gathered.

ELIGIBILITY:
Inclusion Criteria:

* Performance status: Karnofsky score 70 or better or WHO performance status 2 or better
* Diagnosis: Histological, cytological and clinical findings are consistent with squamous cell carcinoma of the head and neck
* Primary tumor diameter as determined clinically or from contrast enhanced CT or T1-weighed MRI scan must be at least 15 mm
* Patients with nodal neck metastases of head and neck cancer are eligible
* Mental status: Patients must be able to understand the meaning of the study
* The patient must sign the appropriate Ethical Committee (EC) approved informed consent documents in the presence of the designated staff
* Patient, if female, must not be pregnant or lactating at the time of the study

Exclusion Criteria:

* Patient must have no history of serious haematologic, cardiovascular, liver or kidney disease.
* Patient must have no history of previous chemotherapy or biological therapy or RT for treatment of head and neck cancer.
* Patient must not have an uncontrolled serious infection
* Patients with organ metastases in liver, bone, brain or lung.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Minn, Professor, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 were recruited, 10 started and completed
Pre-assignment Details: 1 patient withdrawn because of a negative FDG PET scan
Groups:
- 18F-EF5 PET/CT Scan: 18F-EF5
  Pretreatment PET/CT-scan (performed two times)
Period: Overall Study
Arm/Group | 18F-EF5 PET/CT Scan
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 18F-EF5 PET/CT Scan: 10 pts with HNSCC. See Table 1 (p. 163) in Eur J Nucl Med Mol Imaging 2018;45:161-169 https://doi.org/10.1007/s00259-017-3857-3
Arm/Group | 18F-EF5 PET/CT Scan
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Finland | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 18F-EF5 Standardized Uptake Values (SUV)
Description: Standardized Uptake Values (SUV) are determined in the acquisition images of the [18F]EF5 studies.The difference between the baseline and second SUV is calculated and Bland-Altman plots are generated to compare the group means
Time Frame: Baseline and 7 days (ie time between the two scans)
Population: Head and neck squamous cell carcinoma
Measure: Mean (Standard Deviation); unit: SUVmax
Groups:
- Patients With Stage III-IV Head and Neck Cancer: Patients undergoing radiation treatment planning who receive pretreatment PET/CT-scan twice within 1 week as an experimental procedure
Arm/Group | Patients With Stage III-IV Head and Neck Cancer
Number analyzed (Participants) | 10
SUVmax | 1.49 (0.16)

ADVERSE EVENTS:
Arm/Group | 18F-EF5 PET/CT Scan
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No